CLINICAL TRIAL: NCT01273896
Title: A Phase 2 Open-label Study of STA-9090 for Patients With Metastatic Breast Cancer
Brief Title: Open-label Study of STA-9090 for Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-145
Record Dates: First submitted 2011-01-06; First posted 2011-01-11 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: STA-9090; advanced breast cancer; 10-145
MeSH Terms: conditions — Breast Neoplasms | interventions — STA 9090

ARMS (1):
- STA-9090 (Experimental): This will be a monotherapy, open-label phase 2 study of STA-9090 in patients who have metastatic breast cancer.
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090 — All patients will receive 200 mg/m2 of STA-9090 once weekly by a 1-hour IV infusion for three consecutive weeks followed by a 1 week dose-free interval. Subjects tolerating therapy may continue on study until disease progression.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, STA-9090 has on the patient and their breast cancer.

STA-9090 is an experimental drug that works by breaking down cancer proteins. When the cancer proteins are destroyed, the cancer cells die. STA-9090 is an experimental drug that is not yet approved for the treatment of cancer by the United States (FDA) Food and Drug Administration . STA-9090 has been tested in cancer patients in other trials and a safe dose for this drug has been found. We are now interested to see how active this drug is against breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients must be at least 18 years of age
* Pathologically confirmed diagnosis of breast cancer
* Metastatic or advanced stage breast cancer
* Prior treatment with at least one and no more than three lines of biologic and/or chemotherapy for metastatic breast cancer (excluding hormonal therapy)
* Patients with HER2+ disease must have received prior treatment with Trastuzumab
* Patients with ER and/or PR+ disease must have received prior treatment with hormonal therapy
* Off cytotoxic chemotherapy or biologic therapy (excluding Hormonal therapy) ≥ 3 weeks
* Measurable disease by RECIST 1.1
* Central nervous system metastases are permitted if treated and radiographically and clinically stable for at least 4 weeks prior to first dose of STA-9090
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Life expectancy of at least 3 months
* Adequate hematologic function as defined by:
* Absolute neutrophil count ≥1,500 cells/μL
* Platelets ≥100,000/μL
* Hemoglobin ≥ 9.0g/dL
* Adequate hepatic function as defined by:
* Serum bilirubin ≤ 1.5 X upper limit of normal (ULN);
* Adequate renal function as defined by a serum creatinine ≤ 1.5 x ULN
* AST, ALT, and alkaline phosphatase ≤ 3 × ULN except for:
* Patients with hepatic metastases: ALT and AST ≤ 5 × ULN
* Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × ULN
* Patients with Gilbert's disease: serum bilirubin < 5 mg/dL
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Female subjects of childbearing potential and males must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry.

Exclusion Criteria:

* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable disease
* Major surgery within 4 weeks prior to first dose of STA-9090
* Poor peripheral venous access for study drug administration. Study drug administration via indwelling catheters allowed only if the catheter is made of silicone material.
* History of severe (grade 3 or 4) allergic or hypersensitivity reactions to excipients (e.g., Polyethylene glycol [PEG] 300 and Polysorbate 80)
* Baseline QTc > 470 msec
* Ventricular ejection fraction (EF) <50% at baseline
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results in the judgment of the investigator
* Seizure disorder or requirement for seizure medication
* Prior treatment with an HSP90 inhibitor
* persistent adverse events of prior therapies that are > 1 grade 1 in severity
* history of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass surgery
* history of or current uncontrolled dysrhythmias, or requirement for antiarrhythmic medications, or Grade 2 or greater left bundle branch block
* New York Heart Association class II/III/IV congestive heart failure with a history of dyspnea, orthopnea, or edema that requires current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta blockers or diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanu Modi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STA-9090
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | STA-9090
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate using RECIST v 1.1 criteria, defined as PR +CR.using RECIST v 1.1 criteria, defined as Partial response + complete response
Time Frame: Radiological imaging studies to evaluate tumor status will be repeated during the rest week (Days 22 to 28) of every third cycle
Measure: Number; unit: participants
Arm/Group | STA-9090
Number analyzed (Participants) | 20
participants | 20

ADVERSE EVENTS:
Arm/Group | STA-9090
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STA-9090 (N=22)
Cardiac General, other (Cardiac disorders) | 1 (1)
Death not assoc w CTCAE term- Death NOS (General disorders) | 1 (1)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STA-9090 (N=22)
ALT, SGPT (Investigations) | 2 (5)
AST, SGOT (Investigations) | 4 (9)
Alkaline phosphatase (Investigations) | 4 (8)
Amylase (Investigations) | 2 (7)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (4)
CPK (creatine phosphokinase) (Investigations) | 1 (3)
Creatinine (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (7)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (3)
Hemoglobin (Investigations) | 4 (15)
Hypertension (Vascular disorders) | 1 (1)
INR (Investigations) | 2 (6)
Insomnia (Psychiatric disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Lipase (Investigations) | 2 (4)
Lymphopenia (Investigations) | 4 (5)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (2)
Platelets (Investigations) | 1 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes